CLINICAL TRIAL: NCT03716128
Title: Diagnosis of Renal Osteodystrophy in Patients With Reduced Renal Function Can 18F-PET Replace Bone Histomorphometry
Brief Title: Diagnosis of Renal Osteodystrophy in Patients With Reduced Renal Function
Status: Recruiting | Type: Observational
Sponsor: Ditte Hansen (Other)
Collaborators: University of Copenhagen (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor-Investigator, Ditte Hansen, Associate professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: H-17040409
Record Dates: First submitted 2018-09-26; First posted 2018-10-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Renal Osteodystrophy
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bone Biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low turnover bone disease: PTH<150 pg/ml
  Interventions: Diagnostic Test: 18F-PET
- High turnover bone disease: PTH>300 pg/ml
  Interventions: Diagnostic Test: 18F-PET
- Normal renal function: Patients under examination for prostate cancer
  Interventions: Diagnostic Test: 18F-PET

INTERVENTIONS:
Diagnostic Test: 18F-PET — Bone biopsy and 18F-PET
  Other Names: Bone biopsy

SUMMARY:
The aim of the study is to

1. To describe the bone morphology in patients with reduced renal function and high or low parathyroid hormone (PTH) respectively.
2. To investigate if the non-invasive method 18-Fluoride Positron Emission Tomography (18F-PET) can describe the bone turnover and reflect the bone histomorphologic changes
3. To investigate if non-oxidized PTH reflects bone turnover

DETAILED DESCRIPTION:
Patients with reduced renal function and suspected high turnover or low turnover bone disease are recruited.

A bone biopsy and a 18F-PET scan are performed and it is investigated if the 18F-PET can discriminate high turnover from low turnover bone disease

ELIGIBILITY:
Patients with reduced renal function:

Inclusion Criteria:

-≥ 18 years

* estimated Glomerular Filtration Rate (eGFR) ≤ 20 ml/min/1,73m2
* PTH < 150 pg/ml or PTH > 300 pg/ml

Exclusion Criteria:

* ongoing malignancy
* Allergy towards tetracyclin
* Pregnancy

Control Group:

Inclusion Criteria:

-≥ 18 years

* eGFR >= 60 ml/min
* under examination for c prostata
* Prostatic Specific Antigen (PSA) total <40 µg/l

Exclusion:

* Former kidney disease
* ionized calcium or PTH outside normal range
* Known metabolic bone disease
* treatment with anticoagulants
* Disturbed thrombosis and hemostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under investigation for prostate cancer are recruited as bone healthy controls Patients with reduced renal function and suspected high or low bone turnover are recruited for bone biopsy, blood and urin samples and 18F-PET scan
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Can 18F-PET-CT describe bone formation rate? | The bone biopsy and 18F-PET will be performed during two month for each participant
  The ROC curve for 18F uptake by bone measured as bone plasma clearance (ki) to descriminate between high and low bone turnover measured as bone formation rate
Can non-oxidized PTH describe bone formation rate? | Blood sample and bone biopsy will be performed during two month for each participant
  The relation between non-oxidized PTH in ng/L and bone turnover in bone biopsy described as bone formation rate

SECONDARY OUTCOMES:
Can 18F-PET-CT describe mineral apposition rate? | The bone biopsy and 18F-PET will be performed during two month for each participant
  The ROC curve for 18F uptake by bone measured as bone plasma clearance (ki) to descriminate between high and low bone turnover measured as mineral apposition rate
Can non-oxidized PTH describe mineral apposition rate? | Blood sample and bone biopsy will be performed during two month for each participant
  The relation between non-oxidized PTH in ng/L and bone turnover in bone biopsy described as mineral apposition rate

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No